CLINICAL TRIAL: NCT00006227
Title: Phase II Study of Paclitaxel for Ovarian Stromal Tumors as Second-Line Therapy
Brief Title: Paclitaxel in Treating Patients With Ovarian Stromal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0187; NCI-2011-02054 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG #0187; CDR0000068149; GOG-0187; GOG-0187 (Other: NRG Oncology); GOG-0187 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Results first posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Adult Type Ovarian Granulosa Cell Tumor; Ovarian Gynandroblastoma; Ovarian Sertoli-Leydig Cell Tumor; Ovarian Sex Cord Tumor With Annular Tubules; Ovarian Steroid Cell Tumor
MeSH Terms: conditions — Ovarian gynandroblastoma; Sertoli-Leydig Cell Tumor | interventions — Paclitaxel

ARMS (1):
- Treatment (paclitaxel) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Given IV

SUMMARY:
This phase II trial studies the effectiveness of paclitaxel in treating patients who have ovarian stromal cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the probability of clinical response and toxicity of paclitaxel as second-line chemotherapy in measurable disease patients with malignant tumors of the ovarian stroma.

II. To evaluate the value of inhibin for predicting response.

OUTLINE:

Patients receive paclitaxel intravenously (IV) over 3 hours on day 1. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, then every 6 months for three years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with histologically confirmed ovarian stromal tumor (granulosa cell tumor, granulosa cell-theca cell tumor, Sertoli-Leydig cell tumor [androblastoma], steroid [lipid] cell tumor, gynandroblastoma, unclassified sex cord stromal tumor, sex cord tumor with annular tubules)
* Patients must have recurrent stromal tumor having received no more than one prior chemotherapy regimen
* Patients must have measurable disease as defined by Gynecological Oncology Group (GOG) Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* White blood count equal to or greater than 3000/mcl
* Granulocyte count equal to or greater than 1500/mcl
* Platelet count equal to or greater than 100,000/mcl
* Creatinine equal to or less than 2.0 mg%
* Bilirubin less than or equal to 1.5 times normal
* Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 3 times normal
* Patients with a GOG performance grade of 0, 1 or 2
* Patients of child bearing potential must have a negative pregnancy test and must agree to practice an effective means of birth control
* Patients who have met the pre-entry requirements as specified
* Patients must have signed an approved informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion Criteria:

* Patients with GOG performance grade of 3 or 4
* Patients with a prior invasive malignancy (except non-melanoma skin cancer) who have had any evidence of disease within the last 5 years or whose prior malignancy treatment contraindicates the current protocol therapy
* Patients having received more than one prior chemotherapy regimen
* Patients amenable to cure by surgery
* Patients with prior radiation except for those whose recurrent disease is outside the radiation port

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-11-20 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2016-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Van Le, Principal Investigator — NRG Oncology
Locations (98):
- United States (85):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Western Regional CCOP, Phoenix, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Memorial University Medical Center, Savannah, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Union Hospital of Cecil County, Elkton, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Brookview Research Incorporated, Winston-Salem, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - South Carolina Oncology Associates PA, Columbia, South Carolina
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
- Japan (13):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Sapporo Medical College, Sapporo, Chuo-ku
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Iwate Medical University School of Medicine, Morioka, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Kawasaki Medical School, Okayama-Ken, Kurashiki
  - Keio University, Shinjuku-ku, Tokyo
  - National Hospital Organization-Kobe Medical Center, Kobe
  - Shikoku Cancer Center, Matsuyama
  - National Kyushu Cancer Center, Minamiku
  - Jikei University School of Medicine, Minato-ku, Tokyo
  - Kindai University, Osaka, Osaka
  - Tottori University, Tottori

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Paclitaxel)
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paclitaxel)
Number analyzed (Participants) | 31
Age, Customized [Number; unit: participants]
  < 40 | 7
  40-49 | 8
  50-59 | 9
  >= 60 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Probability of Complete Clinical Response
Description: The probability of complete clinical response (i.e. proportion of participants) (assessed using GOG RECIST criteria) of paclitaxel as second line chemotherapy in measurable disease patients with malignant tumors of the ovarian stroma
Time Frame: Up to 5 years
Population: Eligible and evaluable
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment (Paclitaxel)
Number analyzed (Participants) | 31
Percentage of Participants | 3.2 [0.74 to 15.30]

2. Secondary Outcome: Progression-free Survival
Description: Duration of progression free survival (median) (months)
Time Frame: The period from study entry until disease progression, death or date of last contact
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Treatment (Paclitaxel)
Number analyzed (Participants) | 31
Months | 10.0 [6.0 to 19.6]

3. Secondary Outcome: Overall Survival
Description: Duration of overall survival (median) (months)
Time Frame: The observed length of life from entry into the study to death or the date of last contact
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Treatment (Paclitaxel)
Number analyzed (Participants) | 31
Months | 73.6 [63.7 to 112.9]

ADVERSE EVENTS:
Time Frame: For the duration of treatment and follow-up
Description: Adverse events were defined according to CTC v2.0 for the period of protocol activation through March 31, 2010. Beginning on April 1, 2010 adverse events were defined according to CTCAE v4.0.
Arm/Group | Treatment (Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 16/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel) (N=31)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel) (N=31)
Leukopenia (Blood and lymphatic system disorders) | 19
Neutropenia (Blood and lymphatic system disorders) | 21
Anemia (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Investigations) | 6
Allergic reaction (Immune system disorders) | 4
Cardiovascular (Cardiac disorders) | 4
Constitutional (General disorders) | 18
Dermatologic (Skin and subcutaneous tissue disorders) | 22
Gastrointestinal (Gastrointestinal disorders) | 18
Genitourinary (Renal and urinary disorders) | 4
Hepatic (Hepatobiliary disorders) | 5
Infection / fever (Infections and infestations) | 4
Neurologic (Injury, poisoning and procedural complications) | 21
Metabolic (Metabolism and nutrition disorders) | 6
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6
Ocular (Eye disorders) | 6
Pain (General disorders) | 22
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3

LIMITATIONS AND CAVEATS:
The protocol listed an overall study accrual range of 30 to 37, therefore the study achieved this accrual range (n=31). One patient had an indeterminate response for the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less